CLINICAL TRIAL: NCT00549133
Title: Irbesartan Effects on Endothelial Dysfunction in Hypertensive Type II Diabetic Patients Comparing Atenolol
Acronym: IREDIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9130
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Hypertension; Diabetes Mellitus Type 2
Keywords: Microalbuminaria in hypertensive patients with type II diabetes mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irbesartan

SUMMARY:
To show that Irbesartan improves endothelial dysfunction and the procoagulant state which are thought to be the possible mechanisms, inducing a generalized vasculopathy associated with microalbuminuria and vascular events in type II diabetic hypertensive patients

ELIGIBILITY:
Inclusion Criteria:

* non insulin dependent type II manifest diabetes with glycosilated HbA1c levels over %6.5-8
* mild to moderate hypertension stage I and stage II according to ESC-ESH 2003 (140-180 mmHg)

Exclusion Criteria:

* congestive heart failure
* azotemia
* insulin dependent diabetes
* liver insufficiency
* pregnancy
* cancer

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-10; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of irbesartan on nitric oxide (NO), which has key role in the endothelial dysfunction and the development of pressure vasomotor response, compared to standard therapy (atenolol)

SECONDARY OUTCOMES:
Evaluation of the effect of irbesartan on chronic inflammatory process and tendency for procoagulation, associated with endothelial dysfunction, compared to atenolol.

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)